CLINICAL TRIAL: NCT05545202
Title: A Randomized, Comparative, Double-blind Trial of Pentaisomaltose and Dimethyl Sulphoxide for Cryoprotection of Hematopoietic Stem Cells in Subjects With Multiple Myeloma or Malignant Lymphoma With a Need for Autologous Transplantation
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Pharmacosmos A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P-Pentaisomaltose-CRYO-01
Record Dates: First submitted 2022-09-14; First posted 2022-09-19 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Malignant Lymphoma; Multiple Myeloma
MeSH Terms: conditions — Lymphoma; Multiple Myeloma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The subject, trial personnel, and Pharmacosmos personnel will be blinded to the CPA. Blinding will be obtained by shielding the blinded trial personnel from seeing the preparation of the CPA and having unblinded personnel not involved in any trial assessments (efficacy or safety) responsible for randomization, preparation, and accountability of the CPA. The CPA will not be labelled in a way that would reveal the content of the CPA for the blinded personnel or the subject. CPA accountability will be monitored by an unblinded CRA.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A: Pentaisomaltose 16 % (Other): Pentaisomaltose 40 % sterile solution; 40 mL will be transferred to a total volume of 100 mL, so the final concentration is 16 %.
  Interventions: Other: Pentaisomaltose
- B: DMSO 10 % (Active Comparator): Comparator:
  DMSO 99.9 % sterile solution; 10 mL will be transferred to a total volume of 100 mL, so the final concentration is 10 %.
  Interventions: Other: Pentaisomaltose

INTERVENTIONS:
Other: Pentaisomaltose — Each subject will receive 1 or 2 bags with cryopreserved cells according to randomization group.

SUMMARY:
A randomized, comparative, double-blind trial of pentaisomaltose and dimethyl sulphoxide for cryoprotection of hematopoietic stem cells in subjects with multiple myeloma or malignant lymphoma with a need for autologous transplantation

DETAILED DESCRIPTION:
The trial is a randomized, comparative, double-blind trial comparing the efficacy and safety of pentaisomaltose (PentaHibe®, Pharmacosmos A/S, Holbæk; termed PIM in the following) and dimethyl sulphoxide (DMSO), when used for preservation of harvested hematopoietic stem cells. Approximately 150 subjects with a diagnosis of multiple myeloma or malignant lymphoma (a minimum of 30 % of each diagnosis and an equal distribution in each preservation group) and undergoing autologous stem cell transplantation (ASCT) will be included.

The subjects will be randomized 1:1 to receive ASCT preserved in the following cryo-protective agent (CPA):

* A: PIM 16 %
* B: DMSO 10 %

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥ 18 years
* Multiple myeloma or malignant lymphoma diagnosis in which ASCT is indicated according to the standard procedures at the hospital
* Willing to be hospitalized for minimum 24 hours after the ASCT
* Willingness to participate and signing the ICF

Exclusion Criteria:

* Multiple myeloma or lymphoma invasion of the central nervous system
* Previous treatment with ASCT
* Severe infection
* Unsuitable for apheresis
* Unable to provide ≥3 bags with a cell concentration ≥2.0×106 CD34+ cells/kg bodyweight per bag during apheresis
* Pregnant or nursing women. To avoid pregnancy, women of childbearing potential have to use adequate contraception (e.g., intrauterine devices, hormonal contraceptives, or double barrier method) during the whole trial period and up to 1 year after the last ASCT
* Men, even if surgically sterilized, (i.e., status post vasectomy), who do not agree to practice effective barrier contraception during the entire trial period and through 6 months after the last ASCT, or agrees to completely abstain from heterosexual intercourse
* Any other medical condition which, in the opinion of the Investigator, will put the subject's disease management at risk or may result in the subject being unable to comply with the trial requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-04-30 (Estimated); Primary Completion 2025-02-15 (Estimated); Study Completion 2025-02-15 (Estimated)

PRIMARY OUTCOMES:
Engraftment of hematopoietic stem cells | 19 days
  Incidence of subjects with engraftment of hematopoietic stem cells, defined as 2 consecutive measurements with a neutrophil concentration >0.5×109/L within the first 19 days after ASCT
Incidence of subjects with AEs of special interest (limited) | 24 hours after ASCT
  Incidence of subjects with AEs of special interest (limited) occurring within 24 hours after ASCT: headache, nausea, vomiting, bradycardia, or unpleasant odor

SECONDARY OUTCOMES:
Incidence of subjects with AEs of special interest (limited) | 19 days
  Incidence of subjects with AEs of special interest (limited): headache, nausea, vomiting, bradycardia, or unpleasant odor
Time to engraftment of neutrophil cells | 19 days
  • Time to engraftment of neutrophil cells, defined as 2 consecutive measurements with a neutrophil concentration >0.5×109/L within the first 19 days after ASCT